CLINICAL TRIAL: NCT04392986
Title: Effect of Short-term Sunlight Exposure on Blood Pressure and Pulse Rate in Vitamin D3 Insufficient, Prehypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Ji-Young Park, Professor, Korea University Anam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018AN0153
Record Dates: First submitted 2020-05-04; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Sunlight Exposure

STUDY DESIGN:
Intervention Model Description: Single group parallel study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline (No Intervention): Baseline measurement
- Intervention (Experimental): Sunlight intervention
  Interventions: Other: Sunlight exposure

INTERVENTIONS:
Other: Sunlight exposure — The weather was sunny and found suitable for outside activity and sunlight exposure program, with a mean temperature of 27.0-28.5 °C, the humidity of 64-80%, and global solar exposure of 1.28 to 2.99 MJ/m2 during treatment.[15] Participants were asked to lie on the beach for 45 minutes per day between 2 to 3 pm to avoid extreme skin irritation and sunburn from direct sunlight exposure.
  Arms: Intervention

SUMMARY:
A three-period parallel (baseline, treatment, and post-treatment) design clinical research was conducted. All participants visited a clinical trial center of Korea University Anam Hospital for baseline measurement of clinical variables including ABPM and hematologic biomarkers (ACTH, aldosterone, norepinephrine, cortisol, and 25-hydroxyvitamin D3). After the baseline assessment, participants visited 'Cholipo beach' (Taean, Republic of Korea) for 3 nights and 4 days for the intervention (sunlight exposure program). After a week of wash-out period, post-treatment measurement was processed at Korea University Anam Hospital. Participants were prohibited from vigorous physical activity, alcohol drinking, and smoking during the study period. A normal-sodium diet (2800 mg/day)[14], caffeine and smoking restriction was suggested during the whole study period. To control the effect of circadian rhythm on endocrine blood tests and ABPM, we fixed sampling and monitoring start time at 10:00 am. All participants received the same measurements as they did in the baseline measurement during treatment and post-treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* prehypertensive patients
* vitamin D insufficiency
* age 20-45

Exclusion Criteria:

* medical comorbidity other than prehypertension
* participant using medication
* Subjects with a history of cardiovascular, renal, hepatic, gastrointestinal, hematologic, psychological, or gastrointestinal abnormalities, taking any kind of medications

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 24 hours
  24 hour ambulatory blood pressure monitoring
pulse rate | 24 hours

SECONDARY OUTCOMES:
Weight | 3 weeks
  Weight in kilograms
Height | 3 weeks
  Height in meters
Age | 3 weeks
  Age in years
25-hydroxyvitamin D3 | 3 weeks
  ng/mL
Aldosterone | 3 weeks
  ng/mL
Norepinephrine | 3 weeks
  pg/mL
ACTH | 3 weeks
  pg/mL

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea